CLINICAL TRIAL: NCT05571215
Title: The Effect of Combining Pain Neuroscience Education and Transcranial Direct Current Stimulation on Pain Catastrophizing, Kinesiophobia, and Pain in Patients With Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: High Point University (Other)
Responsible Party: Principal Investigator, Cory Alcon, Assistant Professor, High Point University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-FY2022-81
Record Dates: First submitted 2022-08-24; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Chronic Low-back Pain; Catastrophizing Pain; Kinesiophobia
MeSH Terms: conditions — Kinesiophobia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Pilot study - intervention group only
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Combined tDCS and PNE (Experimental): This is a single-arm pilot study used to evaluate the treatment effects of combining pain neuroscience education (PNE) and transcranial direct current stimulation (tDCS). All participants will receive the same Intervention, which includes five sessions of tDCS to the left dorsolateral prefrontal cortex (DLPFC) plus PNE over two weeks.
  Interventions: Device: Transcranial Direct Current Stimulation; Behavioral: Pain Neuroscience Education

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Five sessions of tDCS will be performed following completions of baseline data collection. This will include 3 sessions during week one and 2 sessions in week 2. A tDCS unit (neuroConn Ilmenau, Germany) will be applied to the left DLPFC with participants in the sitting position for a 20 minutes of tDCS. An anodal 2.0 mA current will be applied to each participant, including a 30-second ramp up at the beginning of stimulation and a 30 second ramp down period and the end of stimulation. The left DLPFC (F3 from EEG 10/20 system) will be located using the Beam F3 measurement system. These parameters are consistent with those used in current literature on tDCS for pain. tDCS procedures will be performed by the PI (CA).
Behavioral: Pain Neuroscience Education — Immediately following completion of each tDCS intervention, participants will be given a one-on-one PNE session provided also by the PT (CA), who is a licensed healthcare provider with expertise in delivery of the content. This educational session will last about 30 minutes. Initial sessions will involve discussion and questioning of participants about their own understanding of their pain and this information will be used to subsequently individualize the forthcoming educational sessions. The educational sessions will follow the content of Explain Pain, a patient booklet, and will include information on the neurophysiology of pain, pain as typical process, the transition from acute to chronic pain, neuroplasticity, central sensitization, factors that promote pain chronicity. Information will be presented verbally along with visuals on paper.

SUMMARY:
Recent literature has shown that individuals with persistent chronic pain often exhibit altered cognitive, affective, and sensorimotor behaviors despite a full recovery of peripheral structural injury. Clinically this can be observed via altered pain behaviors (e.g., pain catastrophizing and kinesiophobia) and increased sensitivity to pressure stimuli, each of which are predictive of poorer outcomes. These alterations are believed to have arisen from maladaptive reorganization of brain networks, including cognitive-evaluative and affective networks. Structurally, decreased gray matter in the dorsolateral prefrontal cortex (DLFPC), a key area in the cognitive-affective processing of pain, has been found in those suffering from chronic musculoskeletal pain. The changes are shown to be reversible when the pain is successfully treated and uniquely connected to cognitive-affective behaviors in that as catastrophizing or fear decreases, DLPFC density increases.

Pain science education (PNE), a cognitive-behavioral intervention, has shown promising effects, especially on cognitive- affective behaviors. Non-invasive brain stimulation, such as transcranial direct current stimulation (tDCS), has also been shown to reduce pain and pain-associated behavioral changes in chronic pain. However, the combined effects of these two interventions have not been investigated. It remains unclear if priming the cognitive-affective circuitry that is conceptualized to support PNE with tDCS will augment the behavioral effect of PNE. Therefore, the primary objective of this pilot study is to examine the effects of combining PNE and tDCS on pain catastrophizing, kinesiophobia, and hypersensitivity to pressure stimuli in patients with chronic low back pain (CLBP). We will also examine the influence of PNE and tDCS on cortical network patterns in a subgroup of participants. The results of this pilot study could support the use of tDCS as a priming agent to increase the effect of cognitive-behavioral interventions such as PNE. With success, this intervention could be safely and easily replicated in the clinical setting and provide a novel approach to treating chronic pain more effectively. In addition, the outcomes can further the understanding of more precisely matching specific cortical targets with the desired behavioral therapy

ELIGIBILITY:
Inclusion Criteria:

* Reports chronic low back pain defined as a back pain problem that has persisted at least 3 months and has resulted in pain on at least half the days in the past 6 months
* Age: 18-65 years
* Score >30 on Pain Catastrophizing Scale

Exclusion Criteria:

* History of previous lower back surgery
* Systemic joint disease (e.g. rheumatoid arthritis)
* Evidence of red flags (e.g. fracture, infection, tumor, cauda equina syndrome)
* Cancer
* Neurological disorders
* Neuropathy
* Raynaud's disease
* Pregnancy
* An inability to maintain the testing and treatment positions (i.e. sitting for >30 minutes).
* Exclusion criteria for the tDCS include:
* A history of significant head trauma
* An electrical, magnetic, or mechanical implantation (e.g. cardiac pacemakers or intracerebral vascular
* clip)
* A metal implant in the head or neck areas
* A history of seizures or unexplained loss of consciousness
* An immediate family member with epilepsy
* The use of seizure threshold lowering medicine
* The current abuse of alcohol or drugs
* A history of psychiatric illness requiring medication controls

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Catastrophizing Scale | Completed prior to first intervention session and immediately following final intervention sessions
  The 13-item PCS (0-52) will be used to determine each participant's pain catastrophizing level. Pain catastrophizing is characterized by the tendency to magnify pain stimulus and to feel helpless in the presence of pain. A higher score indicates higher pain catastrophizing level.
Change in Tampa Scale of Kinesiophobia | Completed prior to first intervention session and immediately following final intervention sessions
  . The 17-item TSK (17-68) will be used to determine each participant's level of fear of movement. A higher score indicates higher level of kinesiophobia.
Change in Stroop Color Word Test | Completed prior to first intervention session and immediately following final intervention sessions
  The Stroop Color and Word Test (SCWT) will be used to assess participants ability to inhibit cognitive interference. Cognitive interference occurs when the processing of one stimulus influences the ability to process another feature of the same stimulus.
Change in Numeric Pain Rating Scale | Completed prior to first intervention session and immediately following final intervention sessions
  The NPRS (0-10) will be recorded by the participants rating their current pain on the day of assessment, 0 being no pain and 10 being the worst imaginable pain.

SECONDARY OUTCOMES:
Change in Comprehensive Trail Making | Completed prior to first intervention session and immediately following final intervention sessions
  The Trail making A and B is used to assess participants ability to sustain focus and shift between sets of different stimuli. Part A: Consists of 25 circles numbered from 1 to 25 randomly distributed over a page of letter size paper. The participant is required to connect the circles with a pencil as quickly as possible in numerical sequence beginning with the number 1. Part B: Consists of 25 circles numbered 1 to 13 and lettered A to L, randomly distributed over a page of paper. The participant is required to connect the circles with a pencil as quickly as possible, but alternating between numbers and letters and taking both series in ascending sequence (i.e. 1, A, 2, B, 3, C…)
Change in Coding Test | Completed prior to first intervention session and immediately following final intervention sessions
Change in Pressure Pain Thresholds | Completed prior to first intervention session and immediately following final intervention sessions
  : PPTs will be measured using a pressure algometer (Wagner Instruments, Greenwich, CT) by a research team member. The algometer will be pressed at a steady rate into the most tender point of low back. Participants will indicate when the applied pressure becomes painful (i.e., pain threshold). Three trials will be performed and the last two measurements will be averaged and used for statistical analysis.

OTHER OUTCOMES:
Functional MRI | Completed with 1-2 weeks prior to intervention protocol and within 1 week of completion of the protocol

CONTACTS AND LOCATIONS:
Locations (1):
- High Point University, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alcon C, Zoch C, Luetkenhaus R, Lyman E, Brizzolara K, Goh HT, Wang-Price S. Combined transcranial direct current stimulation and pain neuroscience education for chronic low back pain: a randomized controlled trial. Pain Med. 2025 Feb 1;26(2):90-97. doi: 10.1093/pm/pnae101. PMID 39400579